CLINICAL TRIAL: NCT06032338
Title: EXPérimentation d'Envoi Postal DIrect à Domicile du kiT de dépistage du Cancer Colorectal Sans Commande préalable [Trial of Direct Home Delivery of Colorectal Cancer Screening Kit Without Pre-ordering]
Brief Title: Trial of Direct Home Delivery of Colorectal Cancer Screening Kit Without Pre-ordering
Acronym: EXPEDIT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Caen (Other)
Collaborators: Institut National de la Santé Et de la Recherche Médicale, France (Other Government); Centre Régional de Coordination des Dépistages des Cancers (CRCDC) Centre Val de Loire (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: 2022-A01914-39
Record Dates: First submitted 2023-07-20; First posted 2023-09-13 (Actual); Last update posted 2023-12-22 (Actual); Status verified 2023-07

CONDITIONS: Colorectal Cancer
Keywords: Screening; Participation
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Intervention Model Description: The number of study arms will differ according to age-group:
  * In 50 or 51 yrs age-group, individuals (n=5760 ) will be randomised in 3 groups: C, B1 and B2 (allocation ratio 2:1:1)
  * In the age-group older than 51 yrs, individuals (n=58240) will be randomised in 2 groups: C, and B1 (allocation 1:1) In the main analysis including both age-groups, B1 and B2 arms would be pooled.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control "C" (Other): Usual care : Screening test (Fecal immunochemical test - FIT) delivery and reminders will be carried out in accordance with the Colorectal cancer population-based organised screening program (CRC-PBOSP) specifications at the time of the study.
  This arm is suitable for both the first screening round in 50-51 years old population, and for the subsequent screening rounds.
  Interventions: Other: CRC screening invitation not including the screening test.
- Intervention "B1" (Experimental): FIT mailed at home within the CRC screening invitation without prior information letter.
  This arm is suitable for both the first screening round in 50-51 years old population, and for the subsequent screening rounds.
  Interventions: Other: Mailing of FIT with invitation
- Intervention "B2" (Experimental): FIT mailed at home within the CRC screening invitation with prior information letter.
  This arm is suitable for the first screening round in 50-51 years old population only.
  Interventions: Other: Mailing of FIT with invitation; Other: Information letter before invitation

INTERVENTIONS:
Other: CRC screening invitation not including the screening test. — The invitation to CRC-PBOSP will only contain informations on how to get the screening test.
  Arms: Control "C"
Other: Mailing of FIT with invitation — The invitation to CRC-PBOSP will contain the CRC screening test.
  Arms: Intervention "B1"; Intervention "B2"
Other: Information letter before invitation — An information letter will be sent to future invitees a few weeks before the invitation, to announce the mailing of the CRC screening kit.
  Arms: Intervention "B2"

SUMMARY:
The effect of mailing FIT with the invitation on participation and colonoscopy rates will be evaluated in a randomized controlled trial conducted in the Centre-Val de Loire (CVL) region, involving 64,000 people from the population eligible for colorectal cancer population-based organised screening program (CRC-PBOSP).

In the "C" control group, invitations, test delivery and reminders will be carried out in accordance with the CRC-PBOSP rules at the time of the study.

Intervention group "B" will evaluate two experimental modes of invitation with direct home mailing of the test:

* Method "B1": invitation with test sent to home without prior information letter
* Method "B2": information letter followed by invitation with test sent home, designed to optimize participation by first-time subjects (aged 50-51) invited to the CRC-PBOSP for the first time.

Ancillary studies will focus 1/ on acceptability of this intervention (qualitative study on a few general practitioners, gastroenterologists and invitees), 2/ on social and geographical inequalities of participation on a subsample of individuals included in EXPEDIT study using ecological indices (EDI, SCALE).

ELIGIBILITY:
Inclusion Criteria:

* 50 to 74 years old
* Resident of Centre Val de Loire French area
* Eligible for CRC screening invitation within the biennal CRC-PBOSP during the inclusion period
* Affiliated to the health insurance scheme

Exclusion Criteria:

* CRC screening exclusion criteria notified to CRCDC-CVL in a previous screening round (family or personal history of CRC/adenoma, inflammatory bowel disease)
* Colonoscopy in the previous 5 years)

Subjects refusing data transmission to research team will be excluded from statistical analyses.

Ages: 50 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64000 (Estimated)
Dates: Start 2023-09-14 (Actual); Primary Completion 2025-03-14 (Estimated); Study Completion 2026-11-14 (Estimated)

PRIMARY OUTCOMES:
Participation to CRC screening program | 16 months after the invitation
  Rate of FIT sent to laboratory for analysis within 16 of months of invitation among invitees.
Performance of colonoscopy in FIT positive patients | 6 months after the positive FIT
  Rate of Colonoscopy within 6 months after positive FIT among invitees with a positive FIT

SECONDARY OUTCOMES:
Participation to CRC screening program at 24 months | 24 months after invitation
  Rate of FIT sent to laboratory for analysis within 24 of months of invitation among invitees.
Time to screening participation | 24 months after invitation
  Time to screening participation within 24 months of invitation among invitees
Colonoscopy in FIT positive patients, 12 months after the positive test | 12 months after the positive test
  Rate of Colonoscopy within 12 months after positive FIT among invitees with a positive FIT
Time to colonoscopy (in FIT positive patients) | 12 months after the positive test
  Time from FIT to colonoscopy within 12 months of positive FIT among invitees with a positive FIT
Colonoscopy findings | 12 months after the positive test
  Rate of colorectal cancer or advanced neaplasia in invitees with a positive FIT
Participation to CRC screening program in first invitees (50-51 yrs-old) | 16 months after invitation
  Rate of FIT sent to laboratory for analysis within 16 of months of invitation among first invitees (50-51 yrs-old)
Cost-effectiveness analysis | 24 months
  Costs of CSC-PBOSP from invitation to colonoscopy when necessary

CONTACTS AND LOCATIONS:
Locations (1):
- Crcdc-Cvl, Tours, France

IPD SHARING:
Plan to Share IPD: No